CLINICAL TRIAL: NCT00749827
Title: Exploring the Renoprotective Effects of Fluid Prophylaxis Strategies for Contrast Induced Nephropathy
Brief Title: Renoprotective Effects of Fluid Prophylaxis Strategies for Contrast Induced Nephropathy (CIN)
Acronym: CIN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding received
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Brendan Barrett, Professor of Medicine, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIS-US-0048
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast Induced Nephropathy, fluid prophylaxis
MeSH Terms: interventions — Glucose; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Intravenous sodium bicarbonate (130 mEq/L) in 4.35% dextrose at 3.5 ml/Kg over 1 hour pre-contrast, followed by the same solution intravenously at 1 ml/Kg/hr for 6 hours
  Interventions: Drug: Bicarbonate Hydration
- 2 (Active Comparator): Hypotonic hydration arm. Intravenous 5% dextrose in water at 3.5 ml/Kg over 1 hour pre-contrast followed by 0.9% saline intravenously at 1 ml/Kg/hr for 6 hours.
  Interventions: Drug: Hypotonic hydration

INTERVENTIONS:
Drug: Bicarbonate Hydration — Intravenous sodium bicarbonate (130 mEq/L) in 4.35% dextrose at 3.5 ml/Kg over 1 hour pre-contrast, followed by the same solution intravenously at 1 ml/Kg/hr for 6 hours. In all cases the maximum rate of fluid permitted is that for a body weight of 110 Kg. Intra-vascular low-osmolal or iso-osmolal contrast (according to operator or institution choice) will be used in the minimal dose needed to complete the required imaging.
  Hypotonic hydration arm. Intravenous 5% dextrose in water at 3.5 ml/Kg over 1 hour pre-contrast followed by 0.9% saline intravenously at 1 ml/Kg/hr for 6 hours.
  Other Names: Sodium Bicarbonate(130 mEq/L) in 4.35% dextrose
  Arms: 1
Drug: Hypotonic hydration — Intravenous 5% dextrose in water at 3.5 ml/Kg over 1 hour pre-contrast followed by 0.9% saline intravenously at 1 ml/Kg/hr for 6 hours.
  Other Names: Dextrose(5%) in Water
  Arms: 2

SUMMARY:
Contrast induced nephropathy (CIN) is a term applied to acute renal failure associated with intravascular injection of iodinated contrast agents typically used for cardiac angiography. CIN occurs in about 15% of those who have had cardiac angiography, with dialysis required by about 0.5% of cases. The development of CIN is associated with other adverse outcomes including major adverse cardiovascular events (MACE) and death. The mechanism underlying the association with MACE and death is unclear and it is largely unknown whether measures reducing the frequency or severity of CIN also reduce these associated adverse events.

The cause of CIN in humans is not known, but many preventive therapies have been tested based on our understanding of the mechanism underlying CIN from animal models. Despite multiple studies, no one drug or therapy has been proven to consistently prevent CIN at this time. Prophylactic fluid therapy is uniformly recommended as a component of preventive approaches for CIN. However, the optimal type, dose and duration of fluid therapy remain unclear. Existing studies suggest a role for isotonic saline[3] or bicarbonate[4]. Initial use of hypotonic fluid followed by isotonic fluid might allow a more rapid and sustained increase in tubular fluid flow by suppression of ADH. This should assist in reducing tubular fluid viscosity and the potential for injury by contrast medium.

The aim of this research program is to design and test strategies for the prevention of CIN in patients undergoing elective cardiac angiography or percutaneous coronary intervention (PCI). The primary purpose of this pilot study will be to determine the biological plausibility of using a hypotonic solution for CIN prophylaxis.

Specific Objectives:

Primary

1. To compare the effects of two fluid prophylaxis strategies for CIN on urine output, urine pH, urine composition (urine metabolic profiling), a novel marker of renal injury (NGAL) and urine osmolality Secondary
2. To assess the relative sensitivity of definitions of CIN based on changes in serum creatinine or cystatin C within 72 hours post contrast.
3. To determine the feasibility of a future multicenter randomized trial of a hypotonic fluid prophylaxis strategy for the prevention of radiocontrast nephropathy.

DETAILED DESCRIPTION:
Study Design We propose a pilot randomized trial evaluating the type of fluid chosen for CIN prophylaxis. This study will be conducted at the Health Sciences Centre, St. John's, and the University of Alberta Hospital, Edmonton.

Proposed Interventions:

Bicarbonate hydration arm. Intravenous sodium bicarbonate (130 mEq per L) in 4.35% dextrose at 3.5 ml per Kg over 1 hour pre-contrast, followed by the same solution intravenously at 1 ml/Kg/hr for 6 hours.

Hypotonic hydration arm. Intravenous 5% dextrose in water at 3.5 ml per Kg over 1 hour pre-contrast followed by 0.9% saline intravenously at 1 ml per Kg per hr for 6 hours.

In all cases the maximum rate of fluid permitted is that for a body weight of 110 Kg. Intra-vascular low-osmolal or iso-osmolal contrast (according to operator or institution choice) will be used in the minimal dose needed to complete the required imaging.

Patient population The patient population for this study will be limited to urban dwellers who meet the following inclusion and exclusion criteria. Our rationale for limiting this study to urban dwellers is that blood and urine samples for NGAL need to be frozen at -70 for shipping, therefore these tests will need to be done at the sites of storage and not in peripheral labs.

Duration of Treatment and Follow up Active treatment is limited to the hours while the patient is in the cardiac catheterization laboratory. Patients will be followed up to 7 days post intervention. They will be asked to provide urine and/or blood samples collected at baseline, pre-catheterization, 2 6, 24, and 48-72 hours post-angiography. They will be followed up by telephone at 7 days post intervention to determine if they experienced any adverse events related to the procedure or the intervention.

Measures Baseline Information Baseline measures will include demographic information, comorbidity, location, and indications for cardiac procedure, type of procedure to be performed. Detailed information about the angiographic procedure will be recorded including type and volume of parenteral contrast used. In addition accurate information regarding baseline blood pressure, use of medications (specifically ACE inhibitors, angiotensin receptor blockers, NSAIDS, and diuretics) will be recorded as well as an evaluation of known risk factors for CIN.

Outcome Measures Blood will be collected for measurement of serum creatinine and cystatin C at baseline just prior to fluid administration, and at 6, 24 and 48-72 hours post-angiography. Urine samples for measurement of urine pH, osmolality, electrolytes and creatinine, and NGAL as well as metabolic profiling will be collected on all patients at baseline, pre cardiac catheterization, 6 hours postcardiac catheterization, at the end of the hydration period. As the majority of these patients will not have indwelling urinary catheters, the urine samples will be collected as close to these time points as possible. A table of sample collection timepoints is appended to this application. Assays will be performed on stored samples at a single laboratory to ensure assay standardization between sites. Duration of hospitalization (if any) will be determined by review of records.

Data collection Identification of potential participants is feasible by review of data collected for pre-admission purposes at each site's catheterization laboratory. Study investigators will work collaboratively with the catheterization labs to identify and screen potential participants. Following introduction by clinical staff, potential participants will be approached by study nurses at each site, either on the day of or the day prior to cardiac angiography. The study nurses will obtain consent, collect baseline information and blood and urine specimens, and contact the local investigator for randomization. Once each patient has been randomized the study nurse will arrange for administration of the study therapies and provide the patient with requisitions for follow up blood work. The study investigator will contact the patients either in person if hospitalized or by phone if discharged post procedure and remind them about specimen collections at each time point.

Sample Size This study is exploratory in nature and therefore not powered to a specific endpoint. Previous studies in this area have demonstrated positive results with sample sizes in the order of 50 -100 subjects. We plan to enroll 100 patients in this study.

Statistical Analysis Analysis will be by intention to treat. P values <0.05 will be considered statistically significant. Given that this is a pilot study there will be no interim analysis.

1. Effect of interventions on urinary outcomes The differences between treatment groups will be analyzed using a linear regression model. Estimates and corresponding 95% confidence intervals will be reported. Additional covariates will be explored. Residual, leverage and influence diagnostics will be examined. As metabolic profiling is a relatively new technology patients will serve as their own controls and the results will be reported as paired t tests, describing changes in metabolism associated with radiocontrast administration. Attempts will be made to determine if fluid type influences changes in metabolic profiles by comparing treatment arms using linear regression techniques.
2. Relationship of changes in NGAL to serum creatinine and cystatin C Diagnostic statistics (such as sensitivity, specificity, ROC curve) will also be explored for change in NGAL level at 24 hours using a common definition of CIN as the reference standard (a 44umol/L or 25% rise in serum creatinine at 72 hours post contrast). Additionally, different time points (4 and 48 hours) for NGAL level will be considered.

Data management Dr. Barrett and Dr. Pannu will oversee the data management for this study. Blood and urine will be collected and stored at -70C locally at both participating centers, which each have appropriate storage facilities

ELIGIBILITY:
Inclusion Criteria:

* Booked for cardiac angiography and/or percutaneous coronary intervention
* Pre-existing reduced kidney function (estimated GFR < 60 mls/min/1.73m2 by MDRD equation[18]).
* Minimum age 20 years
* Able to return to the study site for followup blood work.

Exclusion Criteria:

* Estimated GFR < 15 mls/min/1.73m2 by MDRD equation
* Already on dialysis
* Known current acute kidney failure with serum creatinine rise of > 45 mol/L within 24 hours
* Pulmonary edema - current or within 48 hours
* Clinically significant ascites, edema or other fluid overload
* Uncontrolled hypertension (> 165 mmHg systolic, or > 105 mmHg diastolic)
* Unstable patient requiring IV nitroglycerine, or IV fluid or inotropes for BP support
* Emergency angiography
* Planned primary PCI for acute coronary syndrome or myocardial infarction
* Exposure to iodinated radiocontrast within 3 days prior to study
* Prior anaphylactoid reaction to contrast
* Planned administration of N-acetyl-cysteine, dopamine, fenoldopam or mannitol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Serum creatinine, cystatin C,and urine samples for measurement of urine pH, osmolality, electrolytes and creatinine,NGAL and metabolic profiling | SeCr and Cystatin C will be collected at baseline 6hrs, 24, and 48 -72 hrs post cath, urine at baseline, pre-cath, and 6 hours post angiography

CONTACTS AND LOCATIONS:
Overall Officials: Brendan J. Barrett, MD M.Sc., Principal Investigator — Memorial University of Newfoundland
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador

IPD SHARING:
Plan to Share IPD: Undecided